CLINICAL TRIAL: NCT06116786
Title: A Phase 1 Study of JNJ-86974680, an A2a Receptor Antagonist, Administered as Monotherapy and in Combination With Cetrelimab and Radiotherapy for Advanced Non-small Cell Lung Cancer
Brief Title: A Study of JNJ-86974680 in Participants With Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Enterprise Innovation Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 86974680NSC1001; 86974680NSC1001 (Other: Janssen Research & Development, LLC); 2023-506393-12-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: JNJ-86974680+Cetrelimab (Experimental): Participants will receive JNJ-86974680 alone (dose 1, dose 2, dose 3, and dose 4) daily in 4 cohorts and then along with a set dose of cetrelimab.
  Interventions: Drug: JNJ-86974680; Drug: Cetrelimab
- Part 2: JNJ-86974680+Cetrelimab+Radiation Therapy (RT) (Experimental): Part 2 will consist of 3 cohorts (A, B and C) and participants will receive treatment with the selected dose of JNJ-86974680 in combination with cetrelimab from part 1, in conjunction with radiation.
  Interventions: Drug: JNJ-86974680; Drug: Cetrelimab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: JNJ-86974680 — JNJ-86974680 will be administered.
Drug: Cetrelimab — Cetrelimab will be administered.
Radiation: Radiation Therapy — Radiation therapy will be administered.
  Arms: Part 2: JNJ-86974680+Cetrelimab+Radiation Therapy (RT)

SUMMARY:
The purpose of this study is to determine a safe and tolerable dose(s) of JNJ-86974680 for further research in combination with cetrelimab and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with histologically or cytologically confirmed stage IIIB-IV non-small cell lung cancer (NSCLC)
* Part 1: NSCLC with a known actionable genetic mutation (for example, epidermal growth factor receptor [EGFR], anaplastic lymphoma kinase [ALK], c-ros oncogene 1 [ROS1], v-raf murine sarcoma viral oncogene homolog B1 [BRAF]) must have received all approved targeted therapies and have progressed
* Part 2: No targetable mutations (for example, EGFR [epidermal growth factor receptor], ALK [anaplastic lymphoma kinase], ROS1[c-ros oncogene 1], and BRAF [B-Raf proto-oncogene, serine/threonine kinase])
* Part 1 and Cohort A of part 2: Must have been treated with (a) anti-programmed death protein 1 (anti-PD-1) or programmed cell death ligand 1 (PD-L1) therapy and (b) platinum-based chemotherapy
* For Cohort B of Part 2: Previously treated with anti-PD-1/PD-L1 therapy for metastatic disease as the prior line of therapy
* For Cohort C of Part 2: Treatment naïve
* Adequate organ function

Exclusion Criteria:

* Active central nervous system (CNS) disease involvement
* Active autoimmune disease
* Active infection
* History of solid organ or hematologic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2029-06-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years 5 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 2 years 5 months
  The DLTs are specific adverse events and are defined as any of the following: non-hematologic toxicity and hematological toxicity.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-86974680 | Up to 2 years 5 months
  Cmax is defined as maximum observed plasma concentration of JNJ-86974680.
Area Under the Plasma Concentration-time Curve From Time Zero to Time t (AUC0-t) of JNJ-86974680 | Up to 2 years 5 months
  (AUC0-t) is defined as area under the plasma concentration of JNJ-86974680 versus time curve from the time of dose administration to time of last quantifiable concentration (0-t).
Part 2: Overall Response Rate (ORR) | Up to 2 years 5 months
  ORR is defined as the percentage of participants who have a best response of complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST) version (v)1.1, maintained for at least 4 weeks.
Part 2: Complete Response Rate (CRR) | Up to 2 years 5 months
  CRR is defined as the proportion of participants with a best response of CR.
Part 2: Duration of Response (DOR) | Up to 2 years 5 months
  DoR is defined as the time from the date of first initial documentation of a response to the date of first documented evidence of progression of disease according to immunotherapy response evaluation criteria in solid tumors (iRECIST) or death due to any cause, whichever occurs first.
Part 2: Disease Control Rate (DCR) | Up to 2 years 5 months
  DCR is defined as the percentage of participants who achieve a best of response of PR, CR, or stable disease using RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Enterprise Innovation, Inc Clinical Trial, Study Director — Johnson & Johnson Enterprise Innovation Inc.
Locations (15):
- United States (7):
  - City of Hope, Newnan, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Next Virginia, Fairfax, Virginia
- Germany (2):
  - Charite Research Organisation GmbH, Berlin
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
- South Korea (2):
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. I Politecni La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency